CLINICAL TRIAL: NCT01437930
Title: Influence of Intervention With n-3 PUFA-supplemented Products in Moderate Hypertriglyceridemic Patients on Cardiovascular Risk Factors
Brief Title: Intervention With n-3 Polyunsaturated Fatty Acids (PUFA)-Supplemented Products in Moderate Hypertriglyceridemic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Gerhard Jahreis, Proffessor, University of Jena
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H51_11
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2012-03

CONDITIONS: Hypertriglyceridemia
Keywords: n-3 LC-PUFA; hypertriglyceridemic; human; TAG
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- placebo (Placebo Comparator): products (sausage, bread rolls, milk beverage, wafers) enriched with 20g sunflower oil/d
  Interventions: Dietary Supplement: n-3 PUFA

INTERVENTIONS:
Dietary Supplement: n-3 PUFA — products (sausage, bread rolls, milk beverage, wafers) enriched with Intervention a-c): n-3 rich plant oils/powder
  1. linseed oil (20g/d)(PPM, Magdeburg)
  2. echium oil (20g/d) (HARKE Nutrition)
  3. microalgae powder(12g/d)(HARKE Nutrition)

SUMMARY:
The study was performed to investigate the effects of a daily consumption of n-3 PUFA supplemented products (sausage, bread rolls, wafers, milk beverage) on cardiovascular risk factors in hypertriglyceridemic patients.

DETAILED DESCRIPTION:
Recent studies suggest that n-3 LC-PUFA intake might be useful to prevent coronary heart diseases.

As a precondition for participating in this study, the patients were provided information in writing and verbally about the details of the study. Written informed consent was obtained from all volunteers. Before the beginning of the study, all participants were subject to a medical examination by their general practitioners. Sixty hypertriglyceridemic patients (with triacylglyceride (TAG) values ≥ 150 mg/dl or ≥ 1.7 mmol/L) should entered the study.

The placebo-controlled, randomized double-blind cross-over study consists of two investigation periods of 10 weeks, with a ten-week washout period in between. After the washout period the intervention was crossed between the groups and the respective products were consumed for another 10 weeks. Patients in the placebo period receive 60g sausage, 2 bread rolls (2x50g), 2 wafers and one bottle of the milk beverage daily. These products were enriched with sunflower oil (20g/d).

In the intervention period, the products (60g sausage, 2 bread rolls (2x50g), 2 wafers and one bottle of the milk beverage) were enriched with a) 20g linseed oil, b) 20g echium oil, and c)12g microalgae powder. The daily dose of special n-3 fatty acid amounted to a) 10g alpha linolenic acid (ALA), b 2g stearidonic acid (SDA)+6g ALA, or c) 2g docosahexaenoic acid (DHA).

Venous blood is collected at the beginning and at the end of each period.

ELIGIBILITY:
Inclusion Criteria:

* TAG values ≥ 150 mg/dl or ≥ 1.7 mmol/L

Exclusion Criteria:

* Lipid lowering medications
* Glucocorticoids
* Gastrointestinal or metabolic diseases (e.g., diabetes mellitus, hyperthyroidism or hypothyroidism, hypercholesteremic patients with familial previous impacts)
* Daily alcohol abuse
* Taking dietary supplements (e. g., fish oil capsules, vitamin E)
* Known allergies or foodstuff indigestibility

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
blood lipids (total cholesterol, high density lipoprotein (HDL), low density lipoprotein (LDL), TAG) | 10 weeks

SECONDARY OUTCOMES:
blood pressure | 10 weeks
high sensitive C-reactive protein | 10 weeks
oxidised LDL | 10 weeks
lipoprotein a | 10 weeks
  Lipoprotein(a)
vascular cell adhesion molecule | 10 weeks
  vascular cell adhesion molecule
intracellular adhesion molecule | 10 weeks
  intracellular cell adhesion molecule
fatty acid distribution in plasma lipids and erythrocyte membranes | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Friedrich Schiller University, Institute of Nutrition, Jena, Germany

REFERENCES:
- [Derived] Dittrich M, Jahreis G, Bothor K, Drechsel C, Kiehntopf M, Bluher M, Dawczynski C. Benefits of foods supplemented with vegetable oils rich in alpha-linolenic, stearidonic or docosahexaenoic acid in hypertriglyceridemic subjects: a double-blind, randomized, controlled trail. Eur J Nutr. 2015 Sep;54(6):881-93. doi: 10.1007/s00394-014-0764-2. Epub 2014 Sep 13. PMID 25216712